CLINICAL TRIAL: NCT05882331
Title: Extracorporeal Photopheresis as a Possible Therapeutic Approach to Adults With Severe and Critical COVID-19 Non-responsive to Remdesivir, Dexamethasone and Pharmacological Immunomodulation: an Investigational Study
Brief Title: Extracorporeal Photopheresis as a Possible Therapeutic Approach to Adults With Severe and Critical COVID-19
Acronym: COVID-ECP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Del-Pest Central Hospital - National Institute of Hematology and Infectious Diseases (Other)
Responsible Party: Principal Investigator, Bálint Gergely Szabó, Principal Investigator, Del-Pest Central Hospital - National Institute of Hematology and Infectious Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-ECP
Record Dates: First submitted 2023-05-25; First posted 2023-05-31 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Photopheresis

STUDY DESIGN:
Intervention Model Description: ECP is initiated on study inclusion day by Therakos Cellex system, according to manufacturers' instructions. Each patient receives two ECP cycles for 2 weeks, each consisting of two sessions on consecutive days per week (alltogether four sessions), through a peripheral or central venous route. Cycles 1 and 2 are separated by 5 consecutive days. One ECP session takes ~3 hours, and is separated into 4 phases. On priming, the system performes a series of calibrations to ensure proper operation. During collection, 1500 ml of whole blood is processed to collect a concentrated buffy coat containing white blood cells, while other cells and plasma are reinfused. During the photoactive phase, a prescribed dose of 8-methoxypsoralen is added to the buffy coat, which is then circulated through ultraviolet-A photoactivation. During reinfusion phase, treated cells are automatically reinfused to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extracorporeal photopheresis arm (Experimental): Patients will receive extracorporeal photopheresis on this arm, in conjucntion to standard COVID-19 treatments (remdesivir, dexamethasone, IL-6- and/or JAK-inhibition).
  Interventions: Procedure: Extracorporeal photopheresis

INTERVENTIONS:
Procedure: Extracorporeal photopheresis — ECP is initiated on study inclusion day by Therakos Cellex system, according to manufacturers' instructions. Each patient receives two ECP cycles for 2 weeks, each consisting of two sessions on consecutive days per week (alltogether four sessions), through a peripheral or central venous route. Cycles 1 and 2 are separated by 5 consecutive days. One ECP session takes ~3 hours, and is separated into 4 phases. On priming, the system performes a series of calibrations to ensure proper operation. During collection, 1500 ml of whole blood is processed to collect a concentrated buffy coat containing white blood cells, while other cells and plasma are reinfused. During the photoactive phase, a prescribed dose of 8-methoxypsoralen is added to the buffy coat, which is then circulated through ultraviolet-A photoactivation. During reinfusion phase, treated cells are automatically reinfused to the patient.
  Other Names: Therakos Cellex system

SUMMARY:
Optimal approach for adult patients hospitalized with severe and critical COVID-19 non-responsive to antiviral and immunomodulatory drugs is not well established. The study aim is to evaluate feasibility and safety of extracorporeal photopheresis (ECP) in this setting.

DETAILED DESCRIPTION:
A prospective, single-center investigational study is olanned to be performed at a tertiary referral center for COVID-19. Patients with COVID-19 are screened, and severe or critical COVID-19 cases fulfilling pre-defined clinical and biochemical criteria of non-response for >5 days despite remdesivir, dexamethasone and immunomodulation (tocilizumab, baricitinib, ruxolitinib) are consecutively enrolled. After inclusion, two ECP sessions on two consecutive days per week for 2 weeks are applied. Patients are followed up per protocol from study inclusion, and clinical, virological and radiological outcomes are assessed at end-of-treatment (EOT)+28 days.

ELIGIBILITY:
Hospitalized adult (≥18 years at diagnosis) patients with diagnosed COVID-19 of any illness duration are eligible, and screened for inclusion during daily on-site investigator visits. Patients are consecutively enrolled.

Inclusion criteria:

1. severe or critical COVID-19,
2. clinical and biochemical non-response for >5 consecutive days, despite remdesivir, dexamethasone and immunomodulatory therapies (tocilizumab, baricitinib or ruxolitinib), with or without COVID-19 reconvalescent plasmatherapy, in absence of other causes.

Exclusion criteria:

1. pregnancy or breastfeeding,
2. allergy or contraindications to 8-methoxypsoralen,
3. pre-COVID-19 ECP,
4. written informed consent was not obtainable.

Clinical non-response is defined when ≥2 of the following are met, compared to baseline:

1. persistent fever (non-contact tympanal measurement of >38.0°C) for ≥48 hours, despite antipyretics,
2. persistent or failing COVID-19 severity, according to World Health Organization criteria, by ≥1 stratum after ≥48 hours,
3. persistent or failing partial arterial oxygen tension (PaO2) / inspired oxygen fraction (FiO2), by ≥10% after ≥48 hours, despite respiratory support,
4. radiological progression by infiltrate extension on chest computed tomography (CT), by ≥10% after ≥48 hours,
5. novel requirement of invasive mechanical ventilation, as deemed necessary by an intensive care unit (ICU) team.

Biochemical non-response is defined when ≥2 of the following analytes show persistent or increasing levels by ≥20% after ≥48 hours, compared to baseline:

1. serum lactate dehydrogenase (LDH),
2. serum C-reactive protein (CRP),
3. serum ferritin
4. plasma interleukin-6 (IL-6),
5. D-dimer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | All outcomes are assessed at EOT+28 days and compared to data at inclusion.
  Clinical outcomes are all-cause death, invasive mechanical ventilation and ICU admittance requirement.
Virological outcomes | All outcomes are assessed at EOT+28 days and compared to data at inclusion.
  Virological outcomes are respiratory and blood SARS-CoV-2 RT-PCR positivity.
Radiological outcomes | All outcomes are assessed at EOT+28 days and compared to data at inclusion.
  Radiological outcomes are radiological progression/regression or fixed infiltration on chest CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Valyi-Nagy, Prof. Dr., Study Director — South Pest Central Hospital, National Institute of Hematology and Infectious Diseases
Locations (1):
- South Pest Central Hospital, National Institute of Haematology and Infectious Diseases, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, individial patient data will be available to other researchers upon reasonbla request from the principal infestigator.
Supporting Information: CSR
Time Frame: Data will be available after publication of the results in peer-reviewed journals.
Access Criteria: Anonymized, individial patient data will be available to other researchers upon reasonbla request from the principal infestigator.

REFERENCES:
- [Derived] Szabo BG, Remenyi P, Tasnady S, Korozs D, Gopcsa L, Reti M, Varkonyi A, Sinko J, Lakatos B, Szlavik J, Beko G, Bobek I, Valyi-Nagy I. Extracorporeal Photopheresis as a Possible Therapeutic Approach for Adults with Severe and Critical COVID-19 Non-Responsive to Standard Treatment: A Pilot Investigational Study. J Clin Med. 2023 Jul 29;12(15):5000. doi: 10.3390/jcm12155000. PMID 37568402
- See also: Study website — https://tmkk.dpckorhaz.hu/